CLINICAL TRIAL: NCT05297903
Title: Phase II Trial of XmAb20717 in Patients With Advanced Biliary Tract Cancers
Brief Title: XmAb20717 in Advanced Biliary Tract Cancers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 17221; IRB#850515 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2022-02-17; First posted 2022-03-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XmAb20717 (Experimental): Study participants will receive the recommended phase II dose (10mg/kg) of XmAb20717 by intravenous infusion on days 1 and 15 of a 28-day cycle for up to 2 years.
  Interventions: Drug: XmAb20717

INTERVENTIONS:
Drug: XmAb20717 — 10mg/kg IV
  Other Names: ANTI-PD1 × ANTI-CTLA4 BISPECIFIC MONOCLONAL ANTIBODY

SUMMARY:
This is a single-arm, phase II clinical trial to evaluate the efficacy of XmAb20717 in patients with advanced biliary tract cancers who have progressed on, or were intolerant of, a gemcitabine-based chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged > 18 years of age
4. Patient must have advanced biliary tract cancers (BTC) including intrahepatic, perihepatic, or extrahepatic cholangiocarcinoma or gallbladder carcinoma with histologic or cytologic confirmation who have experienced progression, or intolerance of, systemic therapy with a gemcitabine-based regimen.
5. Patients with tumors harboring an FGFR2 fusion, NTRK fusion, or IDH1 mutation must have received molecularly targeted therapy unless contraindicated or refused. Patients without sequencing results for FGFR2 fusions, NTRK fusions, or IDH1 mutations at the time of screening are permitted to enroll in the study. If sequencing results demonstrating FGFR2 fusions, NTRK fusions, or IDH1 mutations become available after patients have enrolled on the study, patients will be informed of the results and available treatment options but may continue study treatment if they are deriving clinical benefit
6. ECOG performance status of 0 or 1.
7. Measurable or evaluable disease as defined by RECIST v. 1.1.
8. Available archival tissue or willingness to undergo biopsy during the screening period; this requirement can be waived if biopsy deemed infeasible or unsafe by the principal investigator.
9. For females of reproductive potential: Must have a negative serum pregnancy test performed within 7 days of first study treatment and must agree to use such a method during study participation and for an additional 3 months after the last study dose of XmAb20717. Reproductive potential is defined in section 8.2.11.
10. For males of reproductive potential with female partners of reproductive potential (per section 8.2.11): Must use of condoms or other methods to ensure effective contraception with partner during the study and for an additional 4 weeks after the end of XmAb20717 administration as outlined in section 8.2.11. Male subjects must agree not to donate sperm from screening through 4 weeks after completion of study
11. Must have adequate organ and hematopoietic function within 14 days of the start of study treatment as defined in Table 1. Labs from cycle 1 day 1 may be used for eligibility.

Exclusion Criteria:

1. Any concurrent condition requiring the continued or anticipated use of systemic steroids beyond physiologic replacement dosing (excluding non-systemic inhaled, topical skin, nasal, and/or ophthalmic corticosteroids). All other systemic corticosteroids above physiologic replacement dosing must be discontinued at least four weeks prior to first study treatment.
2. Treatment with another investigational drug or other intervention within four weeks prior to the first study treatment date.
3. Treatment with trans-arterial liver embolization, hepatic arterial infusion, or radiation doses of > 30 Gy within 4 weeks prior to the first study treatment date
4. Treatment with chemotherapy within 3 weeks prior to the first study treatment date
5. History of permanent discontinuation of a PD-1 or PD-L1 inhibitor therapy due to an immune related adverse event.
6. Prior treatment with a CTLA-4 inhibitor
7. Pregnant or breastfeeding
8. Known allergic reactions to study drug components.
9. Active brain metastases. Patients with brain metastases must have stable neurological status following local therapy (surgery or radiation) for at least four weeks prior to first study treatment and must be off steroids related to the brain metastases.

   for at least two weeks prior to study treatment.
10. Active drug or alcohol use or dependence as documented in the chart that, in the opinion of the investigator, would interfere with adherence to study requirements.
11. Active bacterial, viral, parasitic, or fungal infection requiring IV therapy within 2 weeks of the start of protocol treatment.
12. A secondary primary malignancy that, in the judgment of the investigator, may affect the interpretation of results.
13. Prior organ allograft or allogeneic bone marrow transplantation.
14. A history of, or active, pneumonitis or interstitial lung disease.
15. Active autoimmune disease. Patients with vitiligo, type 1 diabetes mellitus, endocrinopathies manageable by hormone replacement, and psoriasis not requiring systemic treatment are permitted to enroll. Other autoimmune conditions may be allowable at the discretion of the principal investigator.
16. Receipt of a live-virus vaccine within 30 days prior to first dose of study drug (seasonal flu and COVID-19 vaccines are permitted, as long as they do not contain live virus and are not administered within 24 hours of planned administration of XmAb20717)
17. Known human immunodeficiency virus (HIV) infection with CD4+ T-cell (CD4+) counts < 350 cells/μL, or an HIV viral load greater than 400 copies/mL, or a history of an acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within the past 12 months, or who has not been on established antiretroviral therapy (ART) for at least 4 weeks prior to initiation of study drug dosing. (Effective ART is defined as a drug, dosage, and schedule associated with reduction and control of the viral load. HIV positive subjects who do not meet any of these exclusion criteria are eligible.)
18. Any serious or uncontrolled medical or psychiatric disorder that, in the opinion of the investigator, would prevent the patient from providing informed consent, may increase the risk associated with study participation or study drug administration, impair the ability of the patient to receive study protocol therapy, or interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2026-12-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From therapy initiation, assessed at each restaging scan, for up to 24 months
  Proportion of participants with the best response being complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Progression-free survival | From therapy initiation until progression or death, whichever comes first, for up to 60 months
  Time from study enrollment until disease progression or death with censoring for loss to follow up
Overall survival | From therapy initiation until death, for up to 60 months
  Time from study enrollment until death
Objective Response Rate (ORR) in patients that received prior immunotherapy | From therapy initiation, assessed at each restaging scan, for up to 24 months
  Proportion of participants with the best response being complete response (CR) or partial who received prior immunotherapy.
Objective Response Rate (ORR) in patients who did not received prior immunotherapy | From therapy initiation, assessed at each restaging scan, for up to 24 months
  Proportion of participants with the best response being complete response (CR) or partial who did not receive prior immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mark O'Hara, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT05297903/Prot_SAP_001.pdf